CLINICAL TRIAL: NCT00384059
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Pediatric Vaccinations in the United Kingdom
Brief Title: Study to Evaluate a 13-valent Pneumococcal Conjugate Vaccine in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-007
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Results first posted 2012-08-15 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Vaccines, Pneumococcal
MeSH Terms: interventions — diphtheria-tetanus-five component acellular pertussis-inactivated poliomyelitis -Haemophilus influenzae type b conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 13-valent pneumococcal vaccine
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine; Biological: Pediacel; Biological: NeisVac-C; Biological: Menitorix
- 2 (Active Comparator): 7-valent pneumococcal vaccine
  Interventions: Biological: 7vPnC; Biological: Pediacel; Biological: NeisVac-C; Biological: Menitorix

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — Single 0.5 mL dose given at 2, 3, 4, and 12 months of age
  Arms: 1
Biological: 7vPnC — Single 0.5 mL dose given at 2, 3, 4 and 12 months of age
  Arms: 2
Biological: Pediacel — concommitant vaccine, both at arm 1 and at arm 2, at 2 months, 3 months and 4 months of age
Biological: NeisVac-C — concomittant vaccine, both at arm 1 and at arm 2, at 2 months and 4 months of age
Biological: Menitorix — concomitant vaccine, both at arm 1 and at arm 2, at 12 months of age

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate (13vPnC) vaccine compared to Prevenar (7vPnC), when given concomitantly with routine paediatric vaccines in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2 months (42 to 98 days) at the time of enrollment.
2. Available for entire study period and whose parent(s)/legal guardian(s) could be reached by telephone.
3. Healthy infant, as determined by medical history, physical examination, and judgment of the investigator.
4. Parent(s)/legal guardian(s) had to be able to complete all relevant study procedures during study participation.

Exclusion Criteria:

1. Previous vaccination with licensed or investigational pneumococcal vaccine.
2. Previous vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, or meningococcal vaccines.
3. A previous anaphylactic reaction to any vaccine or vaccine-related component.
4. Contraindication to vaccination with Hib conjugate, diphtheria, tetanus, pertussis, polio, pneumococcal conjugate, or meningococcal conjugate vaccines.
5. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
6. Known or suspected immune deficiency or suppression.
7. History of culture-proven invasive disease caused by S pneumoniae, Neisseria meningitidis, or Hib.
8. Major known congenital malformation or serious chronic disorder.
9. Significant neurological disorder or history of seizure, including febrile seizure, or significant stable or evolving disorders, such as cerebral palsy, encephalopathy, hydrocephalus, or other significant disorders. This did not include resolving syndromes due to birth trauma such as Erb palsy.
10. Receipt of blood products or gamma-globulin (including hepatitis B immunoglobulin and monoclonal antibodies; eg, Synagis®).
11. Participation in another investigational trial. Participation in purely observational studies was acceptable.
12. Infant who was a direct descendant (eg, child or grandchild) of the study site personnel.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 286 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For UK/Great Britian, ukmedinfo@wyeth.com
Locations (11):
- United Kingdom (11):
  - Atherstone
  - Bangor
  - Bristol
  - Co Antrim
  - Coventry
  - Ely
  - London
  - Oxford
  - Plymouth
  - Southampton
  - Weston-super-Mare

REFERENCES:
- [Derived] Rodgers GL, Esposito S, Principi N, Gutierrez-Brito M, Diez-Domingo J, Pollard AJ, Snape MD, Martinon-Torres F, Gruber WC, Patterson S, Thompson A, Gurtman A, Paradiso P, Scott DA. Immune response to 13-valent pneumococcal conjugate vaccine with a reduced dosing schedule. Vaccine. 2013 Oct 1;31(42):4765-74. doi: 10.1016/j.vaccine.2013.08.009. Epub 2013 Aug 16. PMID 23965217
- [Derived] Snape MD, Klinger CL, Daniels ED, John TM, Layton H, Rollinson L, Pestridge S, Dymond S, Galiza E, Tansey S, Scott DA, Baker SA, Jones TR, Yu LM, Gruber WC, Emini EA, Faust SN, Finn A, Heath PT, Pollard AJ. Immunogenicity and reactogenicity of a 13-valent-pneumococcal conjugate vaccine administered at 2, 4, and 12 months of age: a double-blind randomized active-controlled trial. Pediatr Infect Dis J. 2010 Dec;29(12):e80-90. doi: 10.1097/inf.0b013e3181faa6be. PMID 21155091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the United Kingdom (UK) from October 2006 to June 2007.
Pre-assignment Details: Participants were enrolled into the study according to inclusion/exclusion criteria without a screening period.
Groups:
- 13vPnC: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and a combined diphtheria, tetanus, five component acellular pertussis (DT5aP), inactivated poliomyelitis (IPV) and haemophilus influenzae type b (Hib) conjugate vaccine (Pediacel) at the 2- and 4-month visits (infant series). Pediacel was administered without study vaccine at 3-month visit. Participants recieved one single 0.5 mL dose of 13vPnC coadministered with Haemophilus Influenzae Type b (Hib) and Meningococcal C Vaccine (Menitorix) at the 12-month visit (toddler dose).
- 7vPnC: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and a combined diphtheria, tetanus, five component acellular pertussis (DT5aP), inactivated poliomyelitis (IPV) and haemophilus influenzae type b (Hib) conjugate vaccine (Pediacel) at the 2- and 4-month visits (infant series). Pediacel was administered without study vaccine at 3-month visit. Participants recieved one single 0.5 mL dose of 7vPnC coadministered with Haemophilus Influenzae Type b (Hib) and Meningococcal C Vaccine (Menitorix) at the 12-month visit (toddler dose).
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 141 | 145
Vaccinated Dose 1 | 139 | 139
Vaccinated Dose 2 | 136 | 135
Completed | 135 | 132
Not Completed | 6 | 13
Not completed — Not consented | 2 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 135 | 132
Completed | 131 | 122
Not Completed | 4 | 10
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Failed to Return | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 131 | 122
Completed | 130 | 120
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Failed to return | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 120 | 118 | 238
Age Continuous [Mean (Standard Deviation); unit: months] | 2.1 (0.3) | 2.1 (0.2) | 2.1 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 57 | 112
  Male | 65 | 61 | 126

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Meningococcal C Serum Bactericidal Assay (SBA) Titer ≥1:8 and Predefined Antibody Levels for Pertussis and Haemophilus Influenzae Type b in 13vPnC Group Relative to 7vPnC Group After the 2-dose Infant Series.
Description: Percentage of participants achieving a meningococcal C SBA serum antibody titer ≥1:8 and predefined antibody threshold levels with the corresponding 95% CI for concomitant antigens polyribosylribitol phosphate (PRP) in haemophilus influenzae type b [Hib](≥0.15 μg/mL or ≥ 1.0 μg/mL), pertussis toxoid [PT], filamentous haemagglutinin, pertactin [FHA], and pertactin (PRN) (≥5 Elisa Units EU/mL) and fimbrial agglutinogens [FIM] (≥2.2 EU/mL) are presented.
Time Frame: One month after infant series dose 2 (5 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate postinfant series antibody concentration to the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 120 | 118
Percentage of participants
  Meningococcal C ≥ 1:8 titer (n=120,118) | 99.2 [95.4 to 100.0] | 99.2 [95.4 to 100.0]
  Hib (PRP) ≥ 0.15 μg/mL (n=114,102) | 96.5 [91.3 to 99.0] | 98.0 [93.1 to 99.8]
  Hib (PRP) ≥ 1.0 μg/mL (n=114,102) | 85.1 [77.2 to 91.1] | 89.2 [81.5 to 94.5]
  Pertussis PT ≥ 5 EU/mL (n=119,112) | 100.0 [96.9 to 100.0] | 100.0 [96.8 to 100.0]
  Pertussis PT ≥ 17 EU/mL (n=119,112) | 96.6 [91.6 to 99.1] | 95.5 [89.9 to 98.5]
  Pertussis FHA ≥ 5 EU/mL (n=119,113) | 100.0 [96.9 to 100.0] | 100.0 [96.8 to 100.0]
  Pertussis FHA ≥ 7.82 EU/mL (n=119,113) | 100.0 [96.9 to 100.0] | 100.0 [96.8 to 100.0]
  Pertussis FHA ≥ 20 EU/mL (n=119,113) | 94.1 [88.3 to 97.6] | 95.6 [90.0 to 98.5]
  Pertussis PRN ≥ 5 EU/mL (n=119,113) | 100.0 [96.9 to 100.0] | 100.0 [96.8 to 100.0]
  Pertussis PRN ≥ 15 EU/mL (n=119,113) | 92.4 [86.1 to 96.5] | 95.6 [90.0 to 98.5]
  Pertussis FIM ≥ 2.2 EU/mL (n=119,113) | 100.0 [96.9 to 100.0] | 97.3 [92.4 to 99.4]
  Pertussis FIM ≥ 5 EU/mL (n=119,113) | 97.5 [92.8 to 99.5] | 96.5 [91.2 to 99.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Meningococcal C the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 titer was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for concomitant antigens was declared if the lower limit of 2-sided 95% CI for the difference between the 2 groups (13vPnC - 7vPnC) > -10%; Difference = 0.0, 95% CI [-3.8 to 3.9]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 0.15 µg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.5, 95% CI [-7.1 to 3.7]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the difference in percentage between the two groups (13vPnC - 7vPnC) at 1.0 µg/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -4.1, 95% CI [-13.4 to 5.1]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Pertussis PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-3.2 to 3.3]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; For Pertussis PT the difference in percentage between the two groups (13vPnC - 7vPnC) at 17 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 1.1, 95% CI [-4.5 to 7.1]
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; For Pertussis FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-3.2 to 3.2]
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; For Pertussis FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 7.82 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-3.2 to 3.2]
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; For Pertussis FHA the difference in percentage between the two groups (13vPnC - 7vPnC) at 20 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -1.5, 95% CI [-7.9 to 4.8]
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; For Pertussis PRN the difference in percentage between the two groups (13vPnC - 7vPnC) at 5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 0.0, 95% CI [-3.2 to 3.2]
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; For Pertussis PRN the difference in percentage between the two groups (13vPnC - 7vPnC) at 15 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = -3.1, 95% CI [-10.0 to 3.4]
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; For Pertussis FIM the difference in percentage between the two groups (13vPnC - 7vPnC) at 2.2 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 2.7, 95% CI [-0.5 to 7.6]
Statistical Analysis 12: Comparison: 13vPnC vs 7vPnC; For Pertussis FIM the difference in percentage between the two groups (13vPnC - 7vPnC) at 5 EU/mL threshold was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference = 1.0, 95% CI [-4.1 to 6.5]

2. Secondary Outcome: Percentage of Participants Achieving an SBA Titer ≥1:8 for Meningococcal C in 13vPnC Group Relative to 7vPnC Group Before and After the Toddler Dose.
Time Frame: one month after the toddler dose (13 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n)= number of participants with a determinate posttoddler dose antibody concentration to the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 13vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C at the 2- and 4-month visits, Pediacel at the 2-, 3-, and 4-month visits.
- 7vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C at the 2- and 4-month visits, Pediacel at the 2-, 3-, and 4-month visits.
- 13vPnC After Toddler Dose; 7vPnC After Toddler Dose: Participants received Menitorix at the 12-month visit.
Arm/Group | 13vPnC Before Toddler Dose | 7vPnC Before Toddler Dose | 13vPnC After Toddler Dose | 7vPnC After Toddler Dose
Number analyzed (Participants) | 102 | 93 | 109 | 98
Percentage of Participants | 44.1 [34.3 to 54.3] | 49.5 [38.9 to 60.0] | 91.7 [84.9 to 96.2] | 91.8 [84.5 to 96.4]
Statistical Analysis 1: Comparison: 13vPnC Before Toddler Dose vs 7vPnC Before Toddler Dose; For Meningococcal C the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 titer was calculated; Test type: Superiority or Other; Difference = -5.3, 95% CI [-19.7 to 8.8]
Statistical Analysis 2: Comparison: 13vPnC After Toddler Dose vs 7vPnC After Toddler Dose; For Meningococcal C the difference in percentage between the two groups (13vPnC - 7vPnC) at 1:8 titer was calculated; Test type: Superiority or Other; Difference = -0.1, 95% CI [-8.0 to 8.1]

3. Secondary Outcome: Percentage of Participants Achieving a Predefined Antibody Level for Haemophilus Influenzae Type b in the 13vPnC Group Relative to the 7vPnC Group After the Toddler Dose.
Time Frame: one month after toddler dose (13 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (N) = number of participants with a determinate posttoddler dose antibody concentration to the given concomitant antigen.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 105 | 96
Percentage of Participants
  Hib (PRP) ≥0.15 μg/mL | 100.0 [96.5 to 100.0] | 100.0 [96.2 to 100.0]
  Hib (PRP)≥1.0 μg/mL | 99.0 [94.8 to 100.0] | 100.0 [96.2 to 100.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; Difference = 0.0, 95% CI [-3.5 to 3.8]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; Difference = -1.0, 95% CI [-5.3 to 2.8]

4. Primary Outcome: Geometric Mean Titer (GMT) of Meningococcal C Antigen as Measured by SBA in 13vPnC Group Relative to 7vPnC Group After the 2-dose Infant Series
Time Frame: one month after infant series dose 2 (5 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations;(N) = number of participants with a determinate antibody concentration/titer for the specified concomitant antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 120 | 118
titer | 306.20 [251.21 to 373.22] | 345.42 [287.91 to 414.41]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Meningococcal C the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — Non-inferiority for the concomitant antigens was declared if the lower bound of the 2-sided, 95% CI for the GMC ratio (13vPnC group/7vPnC group) was >0.5 (2-fold criterion); Ratio = 0.89, 95% CI [0.68 to 1.16]

5. Primary Outcome: Geometric Mean Antibody Concentration of Haemophilus Influenzae Type b (Hib) Polyribosylribitol Phosphate (PRP) as Measured by Enzyme-linked Immunosorbent Assay (ELISA) in 13vPnC Group Relative to 7vPnC Group After the 2-dose Infant Series
Time Frame: one month after infant series dose 2 (5 months of age)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 114 | 102
μg/mL | 3.40 [2.65 to 4.37] | 4.44 [3.50 to 5.63]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.77, 95% CI [0.54 to 1.08]

6. Primary Outcome: Geometric Mean Antibody Concentration of Pertusis Filamentous Haemagglutinin (FHA), Pertussis Toxoid (PT), Pertactin (PRN), and Fimbrial Agglutinogens (FIM) as Measured by ELISA in 13vPnC Group Relative to 7vPnC Group After the 2-dose Infant Series
Time Frame: one month after infant series dose 2 (5 months of age)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 120 | 118
EU/mL
  Pertussis FHA (n=119,113) | 54.74 [48.25 to 373.22] | 55.99 [49.55 to 414.41]
  Pertussis PT (n=119,112) | 66.26 [59.20 to 74.16] | 67.05 [58.75 to 76.52]
  Pertussis PRN (n=119,113) | 61.33 [51.78 to 72.65] | 61.07 [52.31 to 71.30]
  Pertussis FIM (n=119,113) | 21.72 [18.89 to 24.98] | 21.77 [18.54 to 25.56]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Pertussis FHA the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.98, 95% CI [0.82 to 1.16]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; For Pertussis PT the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 0.99, 95% CI [0.83 to 1.17]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; For Pertussis PRN the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.00, 95% CI [0.80 to 1.26]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; For Pertussis FIM the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Ratio = 1.00, 95% CI [0.81 to 1.23]

7. Secondary Outcome: Geometric Mean Antibody Concentration for Haemophilus Influenzae Type b PRP in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose.
Time Frame: one month after toddler dose (13 months of age)
Population: Evaluable immunogenicity (per protocol) population of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (N) = number of participants with a determinate antibody concentration/titer to the specific concomitant antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 105 | 96
μg/mL | 22.22 [17.66 to 27.96] | 19.75 [16.05 to 24.30]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Haemophilus influenzae type b the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ratio = 1.13, 95% CI [0.83 to 1.53]

8. Primary Outcome: Percentage of Participants in the 13vPnC Group Achieving a Serotype-specific IgG Antibody Concentration ≥0.35 µg/mL Measured 1 Month After the 2-dose Infant Series, Before and After the Toddler Dose
Description: Percentages of participants achieving WHO predefined antibody threshold ≥0.35μg/mL along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented.
Time Frame: one month after infant series dose 2 (5 months of age), before and after toddler dose (12 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate igG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- 13vPnC After Infant Series Dose 2; 13vPnC Before Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C at the 2- and 4-month visits, Pediacel at the 2-, 3-, and 4-month visits.
Arm/Group | 13vPnC After Infant Series Dose 2 | 13vPnC Before Toddler Dose | 13vPnC After Toddler Dose
Number analyzed (Participants) | 120 | 120 | 110
Percentage of Participants
  Common Serotypes - Serotype 4 (n=107,89,102) | 95.3 [89.4 to 98.5] | 24.7 [16.2 to 35.0] | 99.0 [94.7 to 100.0]
  Common Serotypes - Serotype 6B (n=107,86,102) | 40.2 [30.8 to 50.1] | 74.4 [63.9 to 83.2] | 98.0 [93.1 to 99.8]
  Common Serotypes - Serotype 9V (n=104,91,101) | 85.6 [77.3 to 91.7] | 44.0 [33.6 to 54.8] | 98.0 [93.0 to 99.8]
  Common Serotypes - Serotype 14 (n=107,88,101) | 92.5 [85.8 to 96.7] | 92.0 [84.3 to 96.7] | 100.0 [96.4 to 100.0]
  Common Serotypes - Serotype 18C (n=111,91,105) | 92.8 [86.3 to 96.8] | 13.2 [7.0 to 21.9] | 97.1 [91.9 to 99.4]
  Common Serotypes - Serotype 19F (n=109,91,104) | 93.6 [87.2 to 97.4] | 67.0 [56.4 to 76.5] | 98.1 [93.2 to 99.8]
  Common Serotypes - Serotype 23F (n=111,89,104) | 66.7 [57.1 to 75.3] | 37.1 [27.1 to 48.0] | 98.1 [93.2 to 99.8]
  Additional Serotypes - Serotype 1 (n=107,88,101) | 97.2 [92.0 to 99.4] | 50.0 [39.1 to 60.9] | 100.0 [96.4 to 100.0]
  Additional Serotypes - Serotype 3 (n=107,87,102) | 86.0 [77.9 to 91.9] | 12.6 [6.5 to 21.5] | 88.2 [80.4 to 93.8]
  Additional Serotypes - Serotype 5 (n=103,88,101) | 89.3 [81.7 to 94.5] | 78.4 [68.4 to 86.5] | 100.0 [96.4 to 100.0]
  Additional Serotypes - Serotype 6A (n=106,86,99) | 79.2 [70.3 to 86.5] | 79.1 [69.0 to 87.1] | 98.0 [92.9 to 99.8]
  Additional Serotypes - Serotype 7F (n=107,91,100) | 94.4 [88.2 to 97.9] | 71.4 [61.0 to 80.4] | 100.0 [96.4 to 100.0]
  Additional Serotypes - Serotype 19A (n=110,91,103) | 92.7 [86.2 to 96.8] | 86.8 [78.1 to 93.0] | 100.0 [96.5 to 100.0]

9. Primary Outcome: Geometric Mean Antibody Concentration in 13vPnC Group After the 2-dose Infant Series, Before and After the Toddler Dose.
Description: Antibody concentration/geometric mean concentration (GMC) as measured by ELISA for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented with corresponding 2-sided 95% CI.
Time Frame: one month after infant series dose 2 (5 months of age) and before and after toddler dose (12 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to protocol requirements, had valid and determinate assay results, and had no other major protocol violations; (n) = number of participants with a determinate antibody concentration for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Groups:
- 13vPnC After Infant Series Dose 2; 13vPnC Before Toddler Dose; 13vPnC After Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C at the 2- and 4-month visits, Pediacel at the 2-, 3-, and 4-month visits, and Menitorix at the 12-month visit.
Arm/Group | 13vPnC After Infant Series Dose 2 | 13vPnC Before Toddler Dose | 13vPnC After Toddler Dose
Number analyzed (Participants) | 120 | 120 | 110
μg/mL
  Common Serotypes - Serotype 4 (n=107,87,87) | 1.37 [1.16 to 1.62] | 0.21 [0.17 to 0.24] | 3.52 [2.91 to 4.26]
  Common Serotypes - Serotype 6B (n=107,85,85) | 0.26 [0.21 to 0.33] | 0.77 [0.60 to 0.99] | 7.67 [5.88 to 10.01]
  Common Serotypes - Serotype 9V (n=104,88,88) | 0.87 [0.72 to 1.05] | 0.29 [0.24 to 0.36] | 2.46 [2.03 to 2.99]
  Common Serotypes - Serotype 14 (n=107,87,87) | 1.83 [1.47 to 2.27] | 1.34 [1.09 to 1.66] | 11.32 [9.27 to 13.83]
  Common Serotypes - Serotype 18C (n=111,91,91) | 1.37 [1.14 to 1.64] | 0.20 [0.17 to 0.23] | 2.14 [1.82 to 2.53]
  Common Serotypes - Serotype 19F (n=109,90,90) | 2.38 [1.88 to 3.01] | 0.60 [0.46 to 0.79] | 7.25 [5.65 to 9.31]
  Common Serotypes - Serotype 23F (n=111,88,88) | 0.53 [0.42 to 0.67] | 0.24 [0.19 to 0.32] | 3.13 [2.59 to 3.78]
  Additional Serotypes - Serotype 1 (n=107,85,85) | 1.69 [1.41 to 2.04] | 0.39 [0.33 to 0.46] | 5.60 [4.60 to 6.82]
  Additional Serotypes - Serotype 3 (n=107,85,85) | 0.63 [0.56 to 0.71] | 0.14 [0.10 to 0.18] | 0.98 [0.78 to 1.22]
  Additional Serotypes - Serotype 5 (n=103,86,86) | 0.95 [0.79 to 1.14] | 0.59 [0.49 to 0.72] | 3.68 [3.04 to 4.45]
  Additional Serotypes - Serotype 6A (n=106,83,83) | 0.86 [0.68 to 1.07] | 0.81 [0.64 to 1.03] | 6.31 [5.06 to 7.87]
  Additional Serotypes - Serotype 7F (n=107,87,87) | 2.14 [1.75 to 2.62] | 0.56 [0.48 to 0.66] | 4.06 [3.42 to 4.83]
  Additional Serotypes - Serotype 19A (n=110,89,89) | 1.90 [1.54 to 2.34] | 1.01 [0.77 to 1.32] | 11.33 [9.29 to 13.83]

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: During the 4-day period after each dose
Population: The safety population included all participants who received at least 1 dose of vaccine; (n)= number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Groups:
- 13vPnC Dose 1: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Pediacel at 2 months of age.
- 7vPnC Dose 1: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Pediacel at 2 months of age.
- 13vPnC Dose 2: Participants received one single 0.5 mL dose of 13vPnC coadministered with NeisVac-C and Pediacel at 4 months of age.
- 7vPnC Dose 2: Participants received one single 0.5 mL dose of 7vPnC coadministered with NeisVac-C and Pediacel at 4 months of age.
- 13vPnC Toddler Dose: Participants received one single 0.5 mL dose of 13vPnC coadministered with Menitorix at 12 months of age.
- 7vPnC Toddler Dose: Participants received one single 0.5 mL dose of 7vPnC coadministered with Menitorix at 12 months of age.
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 139 | 139 | 136 | 135 | 131 | 122
Percentage of Participants
  Tenderness-Any (n=123,127,114,96,87,71) | 44.7 | 43.3 | 42.1 | 40.6 | 44.8 | 50.7
  Tenderness-Significant (n=116,122,97,89,77,58) | 1.7 | 6.6 | 4.1 | 4.5 | 3.9 | 3.4
  Swelling-Any (n=121,126,106,93,83,68) | 24.8 | 29.4 | 30.2 | 34.4 | 30.1 | 39.7
  Swelling-Mild (n=120,125,105,93,82,66) | 21.7 | 27.2 | 28.6 | 29.0 | 28.0 | 34.8
  Swelling-Moderate (n=118,121,98,88,77,60) | 6.8 | 6.6 | 8.2 | 6.8 | 3.9 | 11.7
  Swelling-Severe (n=115,119,96,88,76,57) | 0.0 | 0.0 | 1.0 | 0.0 | 0.0 | 0.0
  Redness-Any (n=122,126,107,99,85,73) | 22.1 | 39.7 | 39.3 | 40.4 | 38.8 | 53.4
  Redness-Mild (n=122,126,106,99,83,71) | 21.3 | 39.7 | 37.7 | 37.4 | 33.7 | 49.3
  Redness-Moderate (n=116,119,98,88,78,61) | 1.7 | 0.0 | 4.1 | 3.4 | 12.8 | 16.4
  Redness-Severe (n=115,119,97,88,76,57) | 0.0 | 0.0 | 2.1 | 0.0 | 0.0 | 0.0

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events
Description: Systemic events (fever ≥ 38 degrees Celsius [C] but ≤ 39 C, fever >39 C but ≤ 40 C, fever > 40 C, decreased appetite, irritability, increased sleep, decreased sleep, use of medication (Meds) to prevent symptoms, and use of medication to treat symptoms) were collected using an electronic diary; percentage of participants with each event was evaluated.
Time Frame: During the 4-day period after each dose
Population: Safety population included all participants who received at least 1 dose of vaccine; (n) = number of participants reporting yes for at least 1 day or no for all days.
Measure: Number; unit: Percentage of Participants
Arm/Group | 13vPnC Dose 1 | 7vPnC Dose 1 | 13vPnC Dose 2 | 7vPnC Dose 2 | 13vPnC Toddler Dose | 7vPnC Toddler Dose
Number analyzed (Participants) | 139 | 139 | 136 | 135 | 131 | 122
Percentage of Participants
  Fever ≥38°C but ≤39°C (n=116,119,96,88,78,61) | 6.0 | 3.4 | 3.1 | 4.5 | 7.7 | 16.4
  Fever >39°C but ≤40°C (n=115,119,95,88,76,58) | 0.9 | 0.0 | 0.0 | 0.0 | 0.0 | 5.2
  Fever >40°C (n=115,119,96,88,76,57) | 0.0 | 0.0 | 2.1 | 0.0 | 0.0 | 0.0
  Decreased appetite (n=120,129,104,98,92,68) | 39.2 | 34.1 | 35.6 | 37.8 | 39.1 | 44.1
  Irritability (n=128,135,117,119,97,80) | 76.6 | 74.1 | 71.8 | 80.7 | 74.2 | 76.3
  Increased sleep (n=129,129,114,109,88,71) | 69.8 | 66.7 | 51.8 | 56.9 | 38.6 | 40.8
  Decreased sleep (n=119,124,98,100,81,67) | 32.8 | 33.9 | 35.7 | 38.0 | 32.1 | 44.8
  Meds to treat symptoms (n=123,128,108,110,85,72) | 43.9 | 40.6 | 50.9 | 54.5 | 49.4 | 58.3
  Meds to prevent symptoms (n=122,124,117,103,92,77) | 49.2 | 40.3 | 48.7 | 50.5 | 52.2 | 67.5

12. Secondary Outcome: Geometric Mean Titer (GMT) of Meningococcal C Antigen as Measured by SBA in 13vPnC Group Relative to 7vPnC Group After the Toddler Dose
Time Frame: one month after toddler dose (13 months of age)
Population: Evaluable immunogenicity (per protocol) population consisting of eligible participants who adhered to the protocol requirements, had valid and determinate assay results, and had no other major protocol violations;(N)= number of participants with a determinate antibody concentration/titer for the specified concomitant antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 109 | 98
titer | 656.11 [445.46 to 966.38] | 771.67 [509.98 to 1167.64]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; For Meningococcal C the GMC ratio (13vPnC/7vPnC) was calculated; Test type: Superiority or Other; Ration = 0.85, 95% CI [0.48 to 1.49]

ADVERSE EVENTS:
Groups:
- 13vPnC Infant Series: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and a combined diphtheria, tetanus, five component acellular pertussis (DT5aP), inactivated poliomyelitis (IPV) and haemophilus influenzae type b (Hib) conjugate vaccine (Pediacel) at the 2- and 4-month visits. Pediacel was administered without study vaccine at 3-month visit.
- 7vPnC Infant Series: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and a combined diphtheria, tetanus, five component acellular pertussis (DT5aP), inactivated poliomyelitis (IPV) and haemophilus influenzae type b (Hib) conjugate vaccine (Pediacel) at the 2- and 4-month visits. Pediacel was administered without study vaccine at 3-month visit.
- 13vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and a combined diphtheria, tetanus, five component acellular pertussis (DT5aP), inactivated poliomyelitis (IPV) and haemophilus influenzae type b (Hib) conjugate vaccine (Pediacel) at the 2- and 4-month visits (assessment at 5 months of age, 1 month after the infant series). Pediacel was administered without study vaccine at 3-month visit.
- 7vPnC Post-Infant Series: Participants received one single 0.5 mL dose of 7-valent pneumococcal conjugate vaccine (7vPnC) coadministered with meningococcal C-tetanus toxoid conjugate vaccine (NeisVac-C) and a combined diphtheria, tetanus, five component acellular pertussis (DT5aP), inactivated poliomyelitis (IPV) and haemophilus influenzae type b (Hib) conjugate vaccine (Pediacel) at the 2- and 4-month visits (assessment at 5 months of age, 1 month after the infant series). Pediacel was administered without study vaccine at 3-month visit.
- 13vPnC Toddler Series: Participants recieved one single 0.5 mL dose of 13vPnC coadministered with Haemophilus Influenzae Type b (Hib) and Meningococcal C Vaccine (Menitorix) at the 12-month visit (toddler dose).
- 7vPnC Toddler Series: Participants recieved one single 0.5 mL dose of 7vPnC coadministered with Haemophilus Influenzae Type b (Hib) and Meningococcal C Vaccine (Menitorix) at the 12-month visit (toddler dose).
- 13vPnC 6-Month Follow-up: Participants recieved one single 0.5 mL dose of 13vPnC coadministered with Haemophilus Influenzae Type b (Hib) & Meningococcal C Vaccine (Menitorix) at the 12-month visit (assessment at 18 months of age, 6 months after the toddler dose).
- 7vPnC 6-Month Follow-up: Participants recieved one single 0.5 mL dose of 7vPnC coadministered with Haemophilus Influenzae Type b (Hib) and Meningococcal C Vaccine (Menitorix) at the 12-month visit(assessment at 18 months of age, 6 months after the toddler dose).
Arm/Group | 13vPnC Infant Series | 7vPnC Infant Series | 13vPnC Post-Infant Series | 7vPnC Post-Infant Series | 13vPnC Toddler Series | 7vPnC Toddler Series | 13vPnC 6-Month Follow-up | 7vPnC 6-Month Follow-up
Serious Adverse Events (participants affected / at risk) | 1/139 | 3/139 | 5/139 | 2/139 | 1/131 | 2/122 | 2/138 | 0/139
Other Adverse Events (participants affected / at risk) | 111/138 | 105/139 | 9/138 | 8/139 | 72/130 | 61/122 | 1/138 | 1/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC Infant Series (N=139) | 7vPnC Infant Series (N=139) | 13vPnC Post-Infant Series (N=139) | 7vPnC Post-Infant Series (N=139) | 13vPnC Toddler Series (N=131) | 7vPnC Toddler Series (N=122) | 13vPnC 6-Month Follow-up (N=138) | 7vPnC 6-Month Follow-up (N=139)
Breath holding (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophaegeal reflux (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tongue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC Infant Series (N=138) | 7vPnC Infant Series (N=139) | 13vPnC Post-Infant Series (N=138) | 7vPnC Post-Infant Series (N=139) | 13vPnC Toddler Series (N=130) | 7vPnC Toddler Series (N=122) | 13vPnC 6-Month Follow-up (N=138) | 7vPnC 6-Month Follow-up (N=139)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangioma (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 7 | 13 | 0 | 0 | 3 | 4 | 0 | 0
Eye discharge (Eye disorders) | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 17 | 0 | 0 | 12 | 13 | 0 | 0
Vomiting (Gastrointestinal disorders) | 19 | 11 | 0 | 0 | 12 | 13 | 0 | 0
Teething (Gastrointestinal disorders) | 11 | 9 | 0 | 0 | 4 | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 9 | 7 | 0 | 0 | 5 | 6 | 0 | 0
Injection site erythema (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site induration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 32 | 26 | 1 | 0 | 11 | 10 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 16 | 19 | 0 | 1 | 4 | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 15 | 14 | 0 | 1 | 9 | 8 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 7 | 4 | 0 | 0 | 8 | 2 | 0 | 0
Varicella (Infections and infestations) | 2 | 8 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 5 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 4 | 2 | 0 | 0 | 2 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Injection site infection (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0 | 0 | 5 | 3 | 0 | 0
Eczema infected (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Rubella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Physical examination abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
High-pitched crying (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Crying (Psychiatric disorders) | 2 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staring (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 16 | 1 | 0 | 10 | 10 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 0 | 0 | 1 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Grunting (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 11 | 5 | 1 | 2 | 1 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 5 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 | 5 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eczema infantile (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Umbilical erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 55/123 | 55/127 | 0/0 | 0/0 | 39/87 | 36/71 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (any)=present at site of vaccination.
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 48/114 | 39/96 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (any)
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 2/116 | 8/122 | 0/0 | 0/0 | 3/77 | 2/58 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant)=present and interfered with limb movement.
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 4/97 | 4/89 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant)
Induration (Any) (Skin and subcutaneous tissue disorders) | 30/121 | 37/126 | 0/0 | 0/0 | 25/83 | 27/68 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (any)=present at site of vaccination.
Induration (Any) (Skin and subcutaneous tissue disorders) | 32/106 | 32/93 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Any)
Induration (Mild) (Skin and subcutaneous tissue disorders) | 26/120 | 34/125 | 0/0 | 0/0 | 23/82 | 23/66 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (mild)=0.5 centimeters (cm) to 2.0 cm.
Induration (Mild) (Skin and subcutaneous tissue disorders) | 30/105 | 27/93 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (Mild)
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 8/118 | 8/121 | 0/0 | 0/0 | 3/77 | 7/60 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (Moderate)=2.5 cm to 7.0 cm.
Induration (Moderate) (Skin and subcutaneous tissue disorders) | 8/98 | 6/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate)
Induration (Severe) (Skin and subcutaneous tissue disorders) | 0/115 | 0/119 | 0/0 | 0/0 | 0/76 | 0/57 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm.
Induration (Severe) (Skin and subcutaneous tissue disorders) | 1/96 | 0/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe)
Erythema (Any) (Skin and subcutaneous tissue disorders) | 27/122 | 50/126 | 0/0 | 0/0 | 33/85 | 39/73 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (any)=present at site of vaccination.
Erythema (Any) (Skin and subcutaneous tissue disorders) | 42/107 | 40/99 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any)
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 26/122 | 50/126 | 0/0 | 0/0 | 28/83 | 35/71 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (mild)=0.5 cm to 2.0 cm.
Erythema (Mild) (Skin and subcutaneous tissue disorders) | 40/106 | 37/99 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild)
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 2/116 | 0/119 | 0/0 | 0/0 | 10/78 | 10/61 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate)=2.5 cm to 7.0 cm.
Erythema (Moderate) (Skin and subcutaneous tissue disorders) | 4/98 | 3/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate)
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 0/115 | 0/119 | 0/0 | 0/0 | 0/76 | 0/57 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm.
Erythema (Severe) (Skin and subcutaneous tissue disorders) | 2/97 | 0/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe)
Fever ≥38°C but ≤39°C (General disorders) | 7/116 | 4/119 | 0/0 | 0/0 | 6/78 | 10/61 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever ≥38 degrees C but ≤39 degrees C
Fever ≥38°C but ≤39°C (General disorders) | 3/96 | 4/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥38 degrees C but ≤39 degrees C
Fever >39°C but ≤40°C (General disorders) | 1/115 | 0/119 | 0/0 | 0/0 | 0/76 | 3/58 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >39 degrees C but ≤40 degrees C
Fever >39°C but ≤40°C (General disorders) | 0/95 | 0/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >39 degrees C but ≤40 degrees
Fever >40°C (General disorders) | 0/115 | 0/119 | 0/0 | 0/0 | 0/76 | 0/57 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Fever >40 degrees C
Fever >40°C (General disorders) | 2/96 | 0/88 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever >40 degrees C
Decreased appetite (General disorders) | 47/120 | 44/129 | 0/0 | 0/0 | 36/92 | 30/68 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 37/104 | 37/98 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Irritability (General disorders) | 98/128 | 100/135 | 0/0 | 0/0 | 72/97 | 61/80 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 84/117 | 96/119 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Increased sleep (General disorders) | 90/129 | 86/129 | 0/0 | 0/0 | 34/88 | 29/71 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 59/114 | 62/109 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Decreased sleep (General disorders) | 39/119 | 42/124 | 0/0 | 0/0 | 26/81 | 30/67 | 0/0 | 0/0 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 35/98 | 38/100 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.